CLINICAL TRIAL: NCT01694940
Title: North American Mitochondrial Disease Consortium Patient Registry and Biorepository (NAMDC)
Acronym: NAMDC
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michio Hirano, MD, Professor of Neurology, Columbia University
Other Study IDs: AAAF4597; U54NS078059 (NIH)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Mitochondrial Disorders; Mitochondrial Genetic Disorders; Mitochondrial Diseases; Disorder of Mitochondrial Respiratory Chain Complexes; Deletion and Duplication of Mitochondrial DNA
Keywords: mitochondrial disorders; Mito Disease; Mitochondria; Mitochondrial disease; Mitochondrial myopathy, encephalopathy, lactic acidosis, and stroke (MELAS) Syndrome; Myoclonic Epilepsy with Ragged Red Fibers (MERRF); Leber Hereditary Optic Neuropathy (LHON); Leigh Syndrome; Neuropathy, ataxia, and retinitis pigmentosa (NARP); Kearns Sayre syndrome; Alpers Huttenlocher; Pearson; Mitochondrial Neurogastrointestinal Encephalopathy (MNGIE); Barth Syndrome; Coenzyme Q (CoQ) Deficiency; Chronic progressive external ophthalmoplegia (CPEO); DAD; Diabetes and Deafness; Encephalopathy; Encephalomyopathy; Familial Bilateral Striatal Necrosis (FBSN); Hepatocerebral Disease; Leukoencephalopathy; Maternally Inherited Leigh Syndrome (MILS); Complex I Deficiency; Complex II Deficiency; Complex III Deficiency; Complex IV Deficiency; Complex V Deficiency; mitochondrial DNA depletion syndrome; mtDNA depletion syndrome
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies; Brain Diseases; Acidosis, Lactic; Stroke; MELAS Syndrome; Syndrome; MERRF Syndrome; Optic Atrophy, Hereditary, Leber; Leigh Disease; Neuropathy ataxia and retinitis pigmentosa; Kearns-Sayre Syndrome; Visceral myopathy familial external ophthalmoplegia; Barth Syndrome; Ophthalmoplegia, Chronic Progressive External; Diabetes Mellitus; Deafness; Leukoencephalopathies; Maternally Inherited Leigh Syndrome; Mitochondrial complex I deficiency; Cytochrome-c Oxidase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any type of tissue sample can be stored in the biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitochondrial Disease Patients: Patients with possible or known mitochondrial disorders. Patients who are known carriers of mitochondrial or nuclear DNA mutations involved in mitochondrial function.

SUMMARY:
The North American Mitochondrial Disease Consortium (NAMDC) maintains a patient contact registry and tissue biorepository for patients with mitochondrial disorders.

DETAILED DESCRIPTION:
Mitochondrial diseases comprise a group of relatively rare (~1 in 5000 adults) but very serious genetic disorders. Mitochondria are often called the "powerhouses of the cell" because they provide the energy our cells need to live. Mitochondria have their own DNA (mtDNA), but they also rely on DNA from the nucleus (nDNA). Mitochondrial diseases are caused by mutations in either mitochondrial or nuclear DNA that result in poorly functioning mitochondria. This can cause a variety of symptoms including muscle weakness, seizures, mental retardation, dementia, hearing loss, blindness, strokes, diabetes, and premature death. Most mitochondrial diseases are progressive, and we are unable to cure most of these diseases with currently available treatments.

Research into mitochondrial diseases has been hampered by the low frequency of these disorders and by under-diagnosis by clinicians. This has hindered patient recruitment for research studies and clinical trials. The North American Mitochondrial Disease Consortium (NAMDC) was established to help surmount these issues. Led jointly by Drs. Michio Hirano and Salvatore DiMauro, NAMDC is a consortium of several clinicians and researchers with an interest in mitochondrial disease research in the United States and Canada.

By creating a mechanism for the sharing of patient samples with researchers, data and patient contact information, NAMDC will make it easier to conduct clinical and basic laboratory research.

Patient information will be shared through the use of the "Patient Data Registry," a specially-designed database, and patient tissue samples will be shared through the use of the "Patient Sample Biorepository", a storage facility in which patient-derived biological samples will be maintained. The Registry and the Biorepository will hopefully accelerate progress in the understanding and treatment of mitochondrial disease.

Patients can enroll at any of the NAMDC member sites. A web-based remote enrollment is also available at www.namdc.org for eligible patients who reside far from any of the NAMDC participating sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with or suspected to have a mitochondrial disorder
* Adult carriers of known mitochondrial DNA mutations
* Patients with laboratory analysis indicative of a mitochondrial disorder.
* Medical information and tissue samples are also accepted from deceased individuals who fulfill the above criteria.

Exclusion Criteria:

* Patients not suspected of having a mitochondrial disorder
* Patients not suspected of carrying a mitochondrial DNA or nuclear DNA mutation that affects mitochondrial function.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known mitochondrial disorders. People at risk of carrying a mitochondrial DNA mutation Patients with abnormal mitochondrial function
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
There is no primary outcome measure for this study | end of study
  This is a registry protocol and therefore there is no primary outcome measure for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Study Director — Columbia University
Locations (17):
- United States (16):
  - University of California San Diego, San Diego, California
  - Lucile Packard Children's Hospital, Stanford, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainsville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Virtual Site (Remote enrollment), New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Case Western Reserve University, Clevland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital and Regional Medical Center, Seattle, Washington
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data is available upon request and approval by the NAMDC Data Use Committee.

REFERENCES:
- See also: Rare Disease Clinical Research Network NAMDC Home Page — https://www1.rarediseasesnetwork.org/cms/NAMDC